CLINICAL TRIAL: NCT02974036
Title: Patient Enablement in Osteoarthritis - a Longitudinal Study on Patient Education Programs in Primary Health Care
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Eva Ekvall-Hansson, Senior lecturer, associate professor, Lund University
Other Study IDs: 782-14
Record Dates: First submitted 2016-08-17; First posted 2016-11-28 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Patient Education as Topic; Osteoarthritis
Keywords: Patient education; Osteoarthritis; Primary health care
MeSH Terms: conditions — Osteoarthritis | interventions — Patient Education as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient education for osteoarthritis: The intervention in the education program consists of three group lessons of about 90 minutes each where information about ethiology, risk factors, treatment and coping strategies concerning OA is included. The first two lessons are held by a physiotherapist and the third by a so-called expert patient that is a person with OA who shares his or her experiences of how to live with the disease. After the intervention patients are able to choose if they want to exercise at home or in a group, supervised by a physiotherapist.
  Interventions: Other: Patient education for osteoarthritis

INTERVENTIONS:
Other: Patient education for osteoarthritis — Group sessions and optional supervised exercise.

SUMMARY:
The overall purpose is to study quality in patient education by means of the patients' self-rated enablement. Specific aims are:

To assess the validity of the patient enablement instrument in relation to self-efficacy and empowerment; To investigate if patient enablement can be effective in identifying which patients would benefit the most from patient education; To study if patient enablement has any relation to self-efficacy, function or self-rated health; To analyze if patient enablement has a causal effect on health care consumption; To evaluate whether patient education is a cost-effective intervention. The project is a longitudinal study, including patients from a patient education programme for osteoarthritis in primary health care. Data consist of patient reported outcome measures and health care consumption. Cost-effectiveness and cost-utility analysis will be used. Inclusion of patients will start August 2016. Analyses of data and manuscript writing will be performed in 2018-2019. Researchers included are from primary health care settings and researchers in the field of OA, patient education and health economy. Our increasingly older and more inactive population will raise huge demands on the health care. The importance of optimizing treatments that are available in primary health care cannot be underestimated. The project will contribute with important knowledge about the patient's own process of getting well.

DETAILED DESCRIPTION:
The project is a longitudinal study, including patients who are referred to patient education for osteoarthritis in primary health care and is planned to follow the patients one year before baseline measures as well as one year after baseline measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are referred to patient education for OA in primary health care
* Speaks and write Swedish

Exclusion Criteria:

* Not having OA
* Not able to speak or write Swedish

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Patient enablement | directly after intervention
  Questionnaire

SECONDARY OUTCOMES:
Arthritis Self Efficacy Scale | before intervention, directly after intervention and at 3 and 9 month follow up
  Questionnaire

OTHER OUTCOMES:
Swedish Rheumatic Empowerment Scale | Before intervention, directly after intervention and at 3 and 9 month follow up
  Questionnaire
EQ5D index | Before intervention, directly after intervention and at 3 and 9 month follow up
  Questionnaire
Health care consumption | 12 months before baseline and 12 months after baseline
  Linked register data from the Skåne Health Care Register
Sick leave | 12 months before baseline and 12 months after baseline
  Linked register data from the Swedish Social Insurance Agency
EQ5D Health barometer | Before intervention, directly after intervention and at 3 and 9 month follow up
  visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ekvall Hansson, Ass prof, Principal Investigator — Lund University
Locations (1):
- Primary Health Care, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hansson EE, Jonsson-Lundgren M, Ronnheden AM, Sorensson E, Bjarnung A, Dahlberg LE. Effect of an education programme for patients with osteoarthritis in primary care--a randomized controlled trial. BMC Musculoskelet Disord. 2010 Oct 25;11:244. doi: 10.1186/1471-2474-11-244. PMID 20969809
- [Derived] Akesson KS, Sunden A, Stigmar K, Eek F, Pawlikowska T, Hansson EE. Empowerment and enablement and their associations with change in health-related quality of life after a supported osteoarthritis self-management programme - a prospective observational study. Arch Physiother. 2023 Sep 22;13(1):18. doi: 10.1186/s40945-023-00172-7. PMID 37735517
- [Derived] Akesson KS, Sunden A, Stigmar K, Fagerstrom C, Pawlikowska T, Ekvall Hansson E. Enablement and empowerment among patients participating in a supported osteoarthritis self-management programme - a prospective observational study. BMC Musculoskelet Disord. 2022 Jun 8;23(1):555. doi: 10.1186/s12891-022-05457-9. PMID 35676666
- See also: BOA registry — https://boa.registercentrum.se/